CLINICAL TRIAL: NCT03009864
Title: The Multi-Center Clinical Study of Tang Shen Prescription on Type 2 Diabetic Kidney Disease in Early Stage
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); Zhengzhou City Hospital of Traditional Chinese Medicine (Other); Shijiazhuang City Hospital of Traditional Chinese Medicine (Unknown); Baoding City Hospital of Traditional Chinese Medicine (Unknown); Hubei Hospital of Traditional Chinese Medicine (Other); Changchun Hospital of Traditional Chinese Medicine (Unknown); Xingtai City Hospital of Traditional Chinese Medicine (Unknown); Medicine Zibo Wanjie Tumor Hospital (Unknown); Zouping Country Hospital of Traditional Chinese Medicine (Unknown); She Country Hospital of Traditional Chinese Medicine (Unknown); Beijing Hospital of TCM (Unknown); Baishi Hospital (Unknown)
Responsible Party: Principal Investigator, Lian-fengmei, Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201507001-11Tangshen
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; TCM; RCT
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tangshen Prescription (Experimental): The prescription contains granules of five Chinese herbal medicines, every bag weighs 4.87g, take it one bag each time, two times a day.
  Interventions: Drug: Tangshen Prescription; Drug: Placebos
- Placebo (Placebo Comparator): Treatment with placebo corresponding to each dose of Tangshen Prescription
  , every bag weighs 4.87g, take it one bag each time, two times a day.
  Interventions: Drug: Tangshen Prescription; Drug: Placebos

INTERVENTIONS:
Drug: Tangshen Prescription — The prescription contains granules of five Chinese herbal medicines, every bag weighs 4.87g, take it one bag each time, two times a day.
Drug: Placebos — Treatment with placebo corresponding to each dose of Tangshen Prescription , every bag weighs 4.87g, take it one bag each time, two times a day.

SUMMARY:
This study is a randomized, double-blinded, placebo-controlled clinical trial on type 2 diabetic Kidney Disease in early stage ( microalbuminuria excretion rate = 20-200mg/min) to evaluate the therapeutic effect of tang shen prescription. 632 participants will be recruited for the study, all of whom had type 2 diabetes, serum creatinine concentrations is normal, and no evidence of non-diabetic renal diseases. The subjects will be randomized to treatment with either tang shen prescription or placebo.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo-controlled clinical trial on type 2 diabetic Kidney Disease in early stage ( microalbuminuria excretion rate = 20-200ug/min) to evaluate the therapeutic effect of tang shen prescription.632 participants will be recruited for the study, all of whom had type 2 diabetes, serum creatinine concentrations is normal, and no evidence of non-diabetic renal diseases. The study will last for 24 weeks. Subjects will be randomly divided into two groups, either tang shen prescription or placebo，and both of them would be performed on a basic treatment which includes diabetes education, diabetic diet, rational control of blood glucose, and losartan at 50 mg daily, study group take tang wang prescription. Measurements of microalbuminuria excretion rate, albumin-to-creatinine ration, glomerular filtration rate (GFR), serum creatinine concentrations will be tested monthly, and quantity of 24h urinary protein per three months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetic Kidney Disease in early stage;
2. Aged 30-70;
3. Signed the informed consent.

Exclusion Criteria:

1. Non-diabetic renal disease, such as gout, essential hypertension, tumors, and chronic kidney disease which may cause proteinuria or microalbuminuria.
2. Cardiovascular disease、hepatopathy、kidney disease and hematopoietic disease et al, the serum transaminase was two times larger than the normal valuet、serum creatinine concentration greater than the upper limit of normal value and psychiatric disease.
3. Women with Pregnancy or prepare for pregnancy or lactating.
4. Degree of renal failure have developed to the stage of hypoxemia and uremia.
5. Patients participate in other clinical researchers within a month.
6. Patients have been treated with the angiotensin receptor blocker (ARB) drugs to treat diabetic kidney disease except for losartan within a month.
7. Patients have been treated with angiotensin-converting enzyme inhibitors (ACEI) drugs to treat diabetic kidney disease within a month.
8. Systolic blood pressure over 160mmHg or diastolic blood pressure over 100mmHg.
9. Patients with diabetic ketosis, ketoacidosis and severe infections within a month.
10. Patients addicting alcohol, psychoactive substances within 5 years.
11. According to the researcher's judgment, there are other diseases or situations that can reduce the possibility of entering the group or complicate the group, such as frequent changes in the working environment and unstable living environment.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-09 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
changes of albumin-to-creatinine ration | 0 week,4 weeks, 8 weeks,12weeks,16weeks, 20weeks, 24weeks

SECONDARY OUTCOMES:
number of participants of diabetic kidney disease in macroalbuminuria stage | 0 week, 4 weeks,8 weeks, 12weeks,16weeks, 20weeks, 24weeks
number of participants whose microalbuminuria excretion rate < 20ug/min | 0 week, 4 weeks, 8 weeks,12weeks,16weeks, 20weeks, 24weeks
change of GFR | 0 week, 4 weeks, 8 weeks,12weeks,16weeks, 20weeks, 24weeks
the rate of doubling the baseline with serum creatinine value | 0 week, 4 weeks, 8 weeks,12weeks,16weeks, 20weeks, 24weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jin D, Huang WJ, Meng X, Yang F, Bao Q, Zhang MZ, Yang YN, Ni Q, Lian FM, Tong XL. Chinese herbal medicine Tangshen Formula treatment for type 2 diabetic kidney disease in the early stage: study protocol for a randomized controlled trial. Trials. 2019 Dec 21;20(1):756. doi: 10.1186/s13063-019-3821-6. PMID 31864393